CLINICAL TRIAL: NCT00119821
Title: Weight Gain Prevention in Hypertensive Smokers
Brief Title: Strategies to Reduce Weight Gain in Hypertensive Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert C. Klesges, Principal Investigator, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 225; R01HL074845 (NIH); NCT00170040 (obsolete NCT alias)
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2011-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity | interventions — Diet, Reducing; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I (Experimental): Behavioral Weight Reduction
  Interventions: Behavioral: Weight Reducing Diet
- II (Other): Exercise
  Interventions: Behavioral: Exercise
- III (Other): Smoking Cessation
  Interventions: Behavioral: Smoking Cessation

INTERVENTIONS:
Behavioral: Weight Reducing Diet — Behavioral intervention
  Arms: I
Behavioral: Exercise — Moderate exercise implemented plus behavioral intervention.
  Arms: II
Behavioral: Smoking Cessation — Nicotine Patch in dosages given based on number of cigarettes per day smoked. 21 mg patch, 14 mg patch, 7 mg patch for total of 6 weeks duration of therapy.
  NRT gum is being provided to assist with relapse prevention. At the randomization visit the participant is given one (1) box of 2mg NRT gum, which consists of (110) pieces. The participant may request up to two (2) more boxes, for a maximum of three (3) boxes per participant.
  Arms: III

SUMMARY:
To evaluate the effectiveness of lifestyle modification following a smoking cessation program in preventing weight gain among hypertensive smokers placed at medical risk by the post-cessation weight gain.

DETAILED DESCRIPTION:
BACKGROUND:

Obesity and smoking are major risk factors for a variety of health-related disorders, such as heart disease, stroke, certain forms of cancer, and diabetes. Recently, it has been reported that up to 65 percent of adults in the United States are overweight or obese. The increasing epidemic of obesity has led to many initiatives to treat obesity and to a number of recent initiatives to prevent weight gain. Similarly, the prevalence of smoking has not declined in the past few years, despite the availability of several clinically and cost-effective smoking cessation programs. One unwanted effect of smoking cessation is weight gain, which, in turn, may exacerbate weight-related health issues. Behavioral programs, and to a lesser degree pharmacological programs, designed to reduce post-cessation weight gain have been successful. However, given that this weight gain is typically cosmetic, it has been determined that such programs should be targeted to those at a higher medical risk as a result of the weight gain (e.g., individuals with hypertension). To our knowledge, no study has evaluated a smoking cessation program, followed by a lifestyle modification program, to prevent weight gain among those placed at medical risk by the post-cessation weight gain, including individuals with hypertension. Some studies find an increased prevalence of hypertension following smoking cessation. It is believed that this is largely (but not solely) due to weight gain following cessation. However, any weight gain in individuals with hypertension places them at risk. Body weight is the single best predictor of adult blood pressure, and blood pressure responds to very small changes in overall body weight.

DESIGN NARRATIVE:

This study will recruit 660 smokers with hypertension or elevated blood pressure. Given that African Americans are at high risk for both post-cessation weight gain and hypertension, the majority of participants recruited will be African American. Participants will be randomly assigned to either of the following: (a) a validated smoking cessation program followed by a validated weight control program (TONE), which consists of changes in dietary intake and physical activity; or (b) the same smoking cessation program followed by a general health education (contact-time control) program. A follow-up evaluation will occur 1 year following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Smoke cigarettes
* Hypertension or elevated blood pressure (a "high normal" designation by the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure [JNC VI] criteria)

Exclusion Criteria:

* Inability to understand consent procedures
* History of an allergic reaction to nicotine replacement therapy
* History of atopic or eczematous dermatitis
* Chronic or severe dermatosis
* History of unstable heart disease, including heart attack, stroke, and unstable angina in the 6 months prior to study entry
* Coronary artery bypass grafting or angioplasty/stent in the 3 months prior to study entry
* Cardiac dysrhythmia (except atrial fibrillation) treated with anti-arrhythmia medication
* History of congestive heart failure (NYHA Class III or IV)
* ECG evidence of 2nd or 3rd degree AV block
* Uncontrolled or stage II hypertension, defined as blood pressure typically greater than 160/100 mm Hg
* History of severe kidney or liver failure
* Current substance abuse (includes alcohol use in excess of 21 drinks a week)
* Severe COPD
* Insulin-dependent diabetes mellitus
* Fasting blood sugar greater than 160 mg/dl
* Hemoglobin less than 11 g/dl
* Untreated hyperthyroidism
* Severe peripheral vascular disease
* Pheochromocytoma
* Pulmonary hypertension
* Valvular heart disease
* Presence of an unstable psychiatric condition
* Current use of a medication that may interfere with study participation or that may increase the risk of side effects from study medication
* Pregnant or plan to become pregnant within the year following study entry
* Planning to move out of the area or travel extensively during the study
* Current medical condition that would preclude any additional changes in diet; dieters and individuals on a special diet will not be excluded from the study
* Unable to modify physical activity, or cannot engage in moderate intensity exercise (e.g., walking); participants who regularly engage in physical activity will not be excluded from the study
* No access to a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2004-09; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Smoking cessation rates | Measured at 1 year
Body weight changes | Measured at 1 year

SECONDARY OUTCOMES:
Changes in dietary intake | Measured at 1 year
Changes in physical activity | Measured at 1 year
Changes in blood pressure and hypertensive status | Measured at 1 year
Changes in blood pressure medication status | Measured at 1 year
Changes in salt intake | Measured at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Klesges, PhD, Study Chair — University of Tennessee Center for Health Sciences